CLINICAL TRIAL: NCT03305211
Title: Biological Collection in Nephrology for the Study of the Links Between Kidney Disease, Immunity System and Cardiovascular Complications
Acronym: NéphroMIC²
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-49
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Kidney Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Intervention Model Description: patients requiring renal biopsy for medical reasons
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological sample (Other): biological sampling will be performed on patients requiring renal biopsy and well-phenotyped patients (diagnosis of renal disease)
  Interventions: Other: sample

INTERVENTIONS:
Other: sample — Participation in NephroMIC involves additional blood samples of 5 tubes (35 mL) and an additional sample of fresh urine.

SUMMARY:
The NephoMIC project is a biological collection in patients of Nephrology, allowing the study of the links between kidney diseases, Immunity system and Cardiovascular complications.

Its aim is to allow the development of a translational research on the theme of "Systemic Nephrology", which concerns both renal complications of autoimmune and inflammatory diseases, and systemic complications of patients with kidney disease, linked to both a state of immunosuppression and an increased risk of cardiovascular complications.

It is based on the proximity between the Clinical investigation Center (CIC) of the hospital, where the samples are received, techniqued and preserved, and the Center of Nephrology and Renal Transplantation of the hospital.

The collection includes blood samples (whole blood, serum, plasma, total blood RNA, PBMC cells), and urine samples (fresh urine).

Participation in the collection is particularly recommended for patients who require a medical renal biopsy in the Nephrology Department. Other well-phenotyped patients (well-defined renal disease diagnosis) may also participate in NephroMIC.

DETAILED DESCRIPTION:
Kidney damage to systemic lupus erythematosus (SLE), anti-cytoplasmic neutrophil cytoplasmic (ANCA) vasculitis or systemic amyloidosis, expose patients to:

* a risk of renal insufficiency, which depends on the severity of the attack, the delay in the initiation of treatment, and the possible occurrence of relapses, which may leave fibrous sequelae and lead to the development of insufficiency chronic renal disease (CKD)
* a risk of immunosuppression and infectious complications, linked to the renal insufficiency itself or to the toxicity of immunosuppressive treatments aimed at controlling renal disease
* an increased risk of cardiovascular complications, linked on the one hand to the activity of the systemic disease and to the endothelial dysfunction it may entail, and on the other hand to the cardiovascular risk associated with the IRC .

Systemic lupus erythematosus (SLE) is a chronic autoimmune disease, evolving in relapses interrupted by periods of remission. Renal impairment of SLE is common (20-30% of patients in Europe) [1] and severe [2], with an impact on patient survival [3] and a risk of progression to chronic renal insufficiency (IRC). Thus, nearly 40% of patients with severe form develop IRC [4], and 5-10% have terminal IRC at 10 years [5,6]. The classification of renal involvement according to the International Society of Nephrology / Renal Pathology Society (ISN / RPS) [7] distinguishes active proliferative forms, requiring immunosuppressive therapy [8], nonproliferative or purely chronic forms. However, renal biopsy remains an invasive procedure [9], which can hardly be repeatedly performed, let alone pre-emptively, although the onset of tissue damage precedes the emergence of clinically detectable proteinuria [10] . In addition, the response of proliferative lupus nephropathy to immunosuppressive therapy is difficult to predict. The progression in treatment is favorable in 70 to 80% of patients with proliferative form, but 20-30% are refractory to the standard treatment, while others retain important chronic lesions leading to chronic renal insufficiency.

There is therefore a crucial need for non-invasive biomarkers to identify lupus patients at risk for developing renal disease and to predict the severity of histological involvement and response to immunosuppressive therapy.

The investigators believe that the pathophysiological complexity of lupus nephropathy can not be summarized to a single biomarker, and that a global "omic" approach could capture this complexity or identify new pathways.

The blood transcriptome study is a non-invasive and usable approach in clinical research, which allowed 10 years ago to identify the signature of lupus interferon (IFN) [11], which had not been detected in serum of patients, and led to new therapeutic pathways. The complexity and size of pan-genomic transcriptomic data may be an obstacle to their analysis and interpretation [12]. Using a modular approach to reduce the size of transcriptomic blood glucose data and facilitate their interpretation, the investigators were able to show the gradation of the interferon signature during lupus [13], and describe the link between neutrophil modular signature and renal impairment of lupus [14].

In addition, the search for noninvasive urinary biomarkers to avoid or limit biopsy indications in the NL, or to predict the response to IS treatment to early adapt the intensity, is of great interest. The current PeptiduLUP study is being conducted to determine the diagnostic and prognostic value of urinary peptidoma analysis during lupus nephropathy. The study of the urinary peptidome could make it possible to refine the indications of renal biopsy in the renal involvement of the lupus.

In addition, there is an increased cardiovascular risk in patients with chronic renal failure (CKD). Our team has demonstrated that the uremic toxins that accumulate in the IRC patients are agonists of the AhR transmission factor and induce endothelial dysfunction with development of a pro-thrombotic [15] and pro-inflammatory phenotype [16] ]. During lupus or vasculitis at ANCA, the risk of cardiovascular complications increases as renal function deteriorates [17,18], while in parallel the risk of immunological outbreak of the disease decreases [19,18]. , 20]. The investigators believe that activation of AhR by uremic toxins may be involved both in increasing the cardiovascular risk of these patients and in inhibiting the autoimmune response.

There is therefore a strong rationale for studying the links between kidney disease, immunity and cardiovascular complications.

The expected results are the identification of new blood (transcriptomic) and urinary (peptidomic) biomarkers for diagnostic and prognostic purposes during renal disease. NephroMIC will also provide research fellowships on biomarkers during renal disease, especially during systemic diseases with renal involvement. The NephroMIC collection will also allow participation in collaborative Nephrology research projects.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient (> 18 years)
* Patient with renal disease
* Patient who signed consent to participate in the study

Exclusion Criteria:

* Pregnant woman
* Severe anemia (Hb <7 g / dL)
* Patient deprived of liberty
* Patient not affiliated to a Social Security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-12-15 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
Blood and urinary biomarkers in renal disease | one day
  biological assay

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique des Hôpitaux de Marseille Hôpital de la Conception, Marseille, France